CLINICAL TRIAL: NCT01832207
Title: Comparison Between Sensory and Motor Transcutaneous Electrical Nervous Stimulation on Electromyographic and Kinesiographic Activity of Patients With Temporomandibular Disorder: a Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Fabrizio Sgolastra, Dr, University of L'Aquila
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMD-224301
Record Dates: First submitted 2013-04-09; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MTS (Active Comparator): Motor threshold of stimulation
  Interventions: Device: Transcutaneous electrical nerve stimulation
- STS (Active Comparator): Sensorial threshold of stimulation
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Placebo (Sham Comparator)
  Interventions: Device: Placebo transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation
  Arms: MTS; STS
Device: Placebo transcutaneous electrical nerve stimulation
  Arms: Placebo

SUMMARY:
Background The purpose of the present controlled clinical trial was to assess the effect of a single 60 min application of transcutaneous electrical nervous stimulation (TENS) at sensory stimulation threshold (STS), compared to the application of motor stimulation threshold (MTS) as well as to untreatment, on the surface electromyographic (sEMG) and kinesiographic activity of patients with temporomandibular disorder (TMD). Methods Sixty female subjects, selected according to the inclusion/exclusion criteria, suffering from unilateral TMD in remission were assigned to MTS, STS or untreatment. Pre- and post-treatment differences in the sEMG activity of temporalis anterior (TA), masseter (MM), digastric (DA) and sternocleidomastoid muscles (SCM), as well in the interocclusal distance (ID), within group were tested using the Wilcoxon test, while differences among groups were assessed by Kruskal-Wallis test; the level of significance was set at p ≤ 0.01.

ELIGIBILITY:
Inclusion Criteria:

* age less than 30 years;
* female gender
* right-handed (7-10 points in Edinburgh inventory);
* presence of complete permanent dentition, with the exception of the third molars;
* normal occlusion;
* diagnosis of unilateral arthrogenous TMD on the Research Diagnostic Criteria for TMD (RDC/TMD), Axis I, groups II and III

Exclusion Criteria:

* having pacemaker or other electrical devices
* previous experience of TENS or biofeedback
* systemic diseases
* history of local or general trauma
* neurological or psychiatric disorders
* muscular diseases
* cervical pain
* bruxism diagnosed by the presence of parafunctional facets and/or anamnesis of parafunctional tooth clenching and/or grinding
* pregnancy
* assumption of anti-inflammatory, analgesic, antidepressant or myorelaxant drugs
* fixed or removable prostheses
* fixed restorations that affected the occlusal surfaces
* previous or concurrent orthodontic or orthognathic treatment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
sEMG values | 60 min

REFERENCES:
- [Derived] Monaco A, Sgolastra F, Pietropaoli D, Giannoni M, Cattaneo R. Comparison between sensory and motor transcutaneous electrical nervous stimulation on electromyographic and kinesiographic activity of patients with temporomandibular disorder: a controlled clinical trial. BMC Musculoskelet Disord. 2013 May 15;14:168. doi: 10.1186/1471-2474-14-168. PMID 23672400